CLINICAL TRIAL: NCT07192939
Title: Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Trial to Evaluate the Efficacy and Safety of HRS-9813 in Subjects With Pulmonary Fibrosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Hengrui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-9813-201
Record Dates: First submitted 2025-09-18; First posted 2025-09-25 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-09

CONDITIONS: IPF and PPF

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group A: HRS-9813 capsules (Experimental)
  Interventions: Drug: HRS-9813 capsules
- Treatment group B: HRS-9813 capsules (Experimental)
  Interventions: Drug: HRS-9813 capsules
- Treatment group C: HRS-9813 capsule mimetic. (Placebo Comparator)
  Interventions: Drug: HRS-9813 capsule mimetic

INTERVENTIONS:
Drug: HRS-9813 capsules — HRS-9813 capsule; High dose
  Arms: Treatment group A: HRS-9813 capsules
Drug: HRS-9813 capsules — HRS-9813 capsule; Low dose
  Arms: Treatment group B: HRS-9813 capsules
Drug: HRS-9813 capsule mimetic — HRS-9813 capsule mimetic
  Arms: Treatment group C: HRS-9813 capsule mimetic.

SUMMARY:
To evaluate the efficacy and safety of HRS-9813 in subjects with pulmonary fibrosis。

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent was obtained to participate in the trial
2. Patients were aged ≥21 years for PPF and ≥45 years for IPF.
3. IPF diagnosed within 7 years before screening (including the screening period) or evidence of progressive ILD within 12 months before screening;
4. HRCT and surgical lung biopsy or transbronchial lung cryobiopsy, when available, support the clinical diagnosis;
5. The central HRCT reading results of PPF at screening showed that the whole lung parenchymal fibrosis was > 10%;
6. Treatment with nintedanib or pirfenidone was discontinued at least 8 weeks before screening or was stabilized for at least 8 weeks;
7. FVC as a percentage of normal predicted value ≥40%;
8. DLCO SB (Hb corrected) as a percentage of normal predicted value ≥25%;
9. Female subjects of childbearing potential must have a negative pregnancy test before the first dose of medication. And must be non-lactating. Female subjects of childbearing potential or male subjects whose partner is a female of childbearing potential agree to be infertile, have a sperm/egg donation plan, and voluntarily use highly effective contraception (including their partner) from the time they sign ICF until 14 days after the last dose of medication, which is the end of safety follow-up.

Exclusion Criteria:

1. IPF cohort: i. Interstitial lung disease (ILD) of other known cause; ii. Diagnosis of sarcoidosis or any systemic autoimmune disease；
2. PPF cohort: IPF diagnosis and UIP features supported by HRCT central reading, surgical lung biopsy, or cryobiopsy pathology.
3. The presence of emphysema of 50% or more on centrally read HRCT or the degree of emphysema greater than the degree of fibrosis on the basis of the most recent HRCT report.
4. The presence of clinically significant nonsubstantial lung disease was considered by the investigator to be likely to affect the assessment of the study.
5. Subjects were known to have pulmonary hypertension requiring treatment with multiple medications.
6. Active tuberculosis infection within 12 months before and/or during screening, or lower respiratory tract infection requiring antibiotic treatment within 4 weeks before and/or during screening, or evidence of active infection on clinical and laboratory tests at the screening/baseline visit.
7. Acute exacerbations of IPF/ILD occurred within 12 weeks before and/or during screening.
8. A history of unstable or worsening cardiac disease within 6 months before screening
9. Uncontrolled atrial or ventricular arrhythmias or the known presence of significant left ventricular dysfunction.
10. A cerebrovascular event leading to hospitalization had occurred within 6 months before screening
11. Had a history of lung volume reduction surgery or transplant, were awaiting lung transplant, or were scheduled to undergo lung volume reduction surgery or transplant during the study period.
12. Subjects with a history of malignancy within the previous 5 years, or a suspicion of malignancy on biopsy, and those for whom the possibility of malignancy could not be reasonably ruled out after additional clinical, laboratory, or other diagnostic evaluation were screened.
13. The patients were positive for hepatitis B surface antigen (HBsAg) or hepatitis C virus antibody (HCVAb) at the time of screening. A test for antibodies to the human immunodeficiency virus (HIV) was not negative at screening.
14. A history of smoking (including e-cigarettes) within 3 months before screening or an unwillingness to quit smoking during the study.
15. Regular alcohol consumption in the 6 months before screening or an unwillingness to reduce alcohol consumption to less than 21 units during the study.
16. He had a history of substance abuse within 6 months before screening.
17. Pregnant or breastfeeding.
18. Treatment with prednisone at a dose of more than 15 mg per day or another systemic glucocorticoid at the equivalent dose was received within 4 weeks before screening and during the study.
19. Use of an IL-6 inhibitor within 3 months before screening and planned use during the study.
20. Disease-modifying antirheumatic drugs or a change in dose were initiated within 3 months before screening.
21. Initiation of mycophenolate mofetil, mycophenolic acid, azathioprine, tacrolimus, methotrexate, leflunomide, or a change in the dose of the above drugs within 3 months before screening; Immunosuppressive drugs could not be started during the treatment phase.
22. Rituximab was used 6 months before screening and was planned for the duration of the study.
23. Participants who had used a potent inhibitor or inducer of cytochrome P450(CYP)3A4 within 4 weeks before randomization or who had to be treated with or planned to be treated with a drug ban during the study.
24. Persons who had participated in a clinical trial of any drug or device within 1 month before screening and who had expected legacy effects of the trial treatment (at the discretion of the investigator) or who were within the follow-up period of a clinical study or the five half-lives of the trial drug before screening.
25. Major surgery (surgery under general anesthesia) that was performed within 3 months before screening or that was planned during the study that, as assessed by the investigator, would affect the determination of the end points.
26. Uncontrolled hypertension was present before screening or randomization.
27. Patients with orthostatic intolerance, orthostatic hypotension, or orthostatic tachycardia, as well as patients with a previous history of these conditions, at screening or before randomization.
28. A history of persistent or active syncope after urination/defecation, a previous known history of syncope, or a concomitant medical condition that increases the risk of syncope.
29. Bilirubin, transaminase, blood routine and other abnormalities exceed the requirements during screening.
30. An electrocardiogram showed a heart rate of less than 55 beats per minute before screening or randomization or a QT interval of at least 500 msec or a QTcF interval of at least 450 msec before randomization.
31. Allergy to drugs in the same class or to any component of HRS-9813.
32. Other reasons for not participating in the study as judged by the investigator.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2025-10-29 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
FVC as a percentage of the predicted value | The baseline period lasted until 26weeks after administration

SECONDARY OUTCOMES:
The rate of change in ppFVC | The baseline period lasted until 26 weeks after administration
Absolute change in FVC. | The baseline period lasted until 26 weeks after administration
Changes in lung carbon monoxide diffusion capacity (DLCO SB) (hemoglobin corrected) and its percentage of the predicted value (ppDLCO SB) (hemoglobin corrected). | The baseline period lasted until 26 weeks after administration
Proportion of subjects with an absolute decline in ppFVC (%) of ≥10% from baseline. | The baseline period lasted until 26 weeks after administration
Proportion of subjects with acute exacerbation of pulmonary fibrosis. | The baseline period lasted until 26 weeks after administration
Proportion of subjects with respiratory-related hospitalizations. | The baseline period lasted until 26 weeks after administration
Proportion of subjects with pulmonary fibrosis-related hospitalizations. | The baseline period lasted until 26 weeks after administration
All-cause mortality. | The baseline period lasted until 26 weeks after administration
Proportion of subjects with pulmonary fibrosis disease progression. | The baseline period lasted until 26 weeks after administration
The changes of the scores of each sub-item and the impact part of the Pulmonary fibrosis questionnaire (L-PF) were observed. | The baseline period lasted until 26 weeks after administration

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Sciences & Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided